CLINICAL TRIAL: NCT01589198
Title: Identification of Molecular Biomarkers to Stratify Patients With Refractory Asthma
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NJH HS-2639
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and lung samples will be retained for RNA purposes.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn more about asthma in people who are not well-controlled with current asthma medication (refractory asthma). The investigators will compare data from refractory asthmatic patients here at National Jewish Health to mild asthmatics subjects and to people without asthma. Study experiments involve looking at samples from all 3 groups and comparing them at a molecular level. These laboratory experiments may help identify subtypes of refractory asthmatics that require different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Able to receive Informed Consent
* At least 18 years of age
* ICS < 880 mcg (FP equivalents)
* PC20<=16 mg/mL
* No more than 1 oral steroid bursts in previous 12 months
* Less that 3 urgent care visit in previous 12 months
* No deterioration with <=25% decrease in steroids
* No near fatal asthma event

Exclusion Criteria:

* Pregnancy
* Current smoker, smoking within the past year or pack/year history >10 years
* Respiratory infection within past 6 weeks
* Antibiotics within the past 6 weeks
* Active lung disease other than asthma
* Cancer within past 5 years (excluding basal cell skin cancer)
* Active or chronic infection
* Hematological or autoimmune disease
* Unable to safely undergo bronchoscopy as determined by doctor or study doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are looking for mild non-smoking asthmatic adults who are well-controlled with their asthma therapy (non-refractory asthmatics).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Determining phenotypes non-invasively | October, 2015
  Comparing invasive phenotyping to non-invasive

CONTACTS AND LOCATIONS:
Overall Officials: Richard Martin, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States